CLINICAL TRIAL: NCT02563899
Title: A Phase 2a Study to Evaluate the Pharmacokinetic, Safety, Tolerability and Clinical Effect of Topically Applied Umeclidinium/GSK573719 in Subjects With Primary Axillary Hyperhidrosis
Brief Title: Pharmacokinetic, Safety, Tolerability, and Clinical Effect of Topical Umeclidinium in Primary Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202093
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Hyperhidrosis
Keywords: Primary Axillary Hyperhidrosis; GSK573719; Hyperhidrosis Disease Severity Scale (HDSS); Topical; PRO; Hyperhidrosis Symptom Severity Measure (HSSM); Umeclidinium
MeSH Terms: conditions — Hyperhidrosis | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium (Experimental): Subjects will receive umeclidinium once daily before bedtime for 14 days.
  Interventions: Drug: Umeclidinium
- Vehicle (Placebo Comparator): Subjects will receive vehicle once daily before bedtime for 14 days.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Umeclidinium — Umeclidinium (GSK573719) 1.85% will be supplied as a clear, colorless solution, free from visible particulates, for topical application. This formulation will be available at a concentration of 18.5 milligrams (mg) umeclidinium parent per gram. 2 mg of this formulation will be applied per square centimeter of the axilla, once a day at night before going to bed for 14 days. The total amount of formulation applied daily to both axillae is expected to range between approximately 204 and 680 mg. Total daily dosage of the active pharmaceutical ingredient (umeclidinium parent) to both axillae will range between approximately 3.8 and 12.6 mg. If certain pre-specified criteria for safety and tolerability are met, consideration will be given to decreasing the dose by decreasing the concentration of the topical formulation to 1.15% for the remaining subjects. This lower strength formulation will contain 11.5 mg parent per gram.
  Arms: Umeclidinium
Drug: Vehicle — The vehicle will be supplied as a clear, colorless solution, free from visible particulates, for topical application. This formulation will be similar to the umeclidinium formulation except that it will be devoid of the umeclidinium parent. 2 mg of the vehicle will be applied per square centimeter of the axilla, once a day at night before going to bed for 14 days. The total amount of vehicle applied daily to both axillae is expected to range between approximately 204 and 680 mg.
  Arms: Vehicle

SUMMARY:
This is a double blind (sponsor unblind), repeat dose, randomized, parallel group, placebo controlled study to assess the pharmacokinetic parameters, safety, tolerability, and clinical effect of topically applied umeclidinium following once daily topical administration to axilla for 14 days in subjects with primary axillary hyperhidrosis. This study will determine whether topically applied umeclidinium can decrease hyperhidrosis without systemic anticholinergic effects (ie. in the range or lower to those obtained after inhaled route) at the highest possible concentration.

Subjects will be dosed by site staff each night immediately before bedtime for 14 days. Subjects will complete gravimetric and Hyperhidrosis Disease Severity Scale (HDSS) measurements, patient reported outcomes (PRO), safety assessments, and/or pharmacokinetic sampling. Follow up visits will occur on days 15, 16, 19, 23 and 28. The total duration of the study will be approximately 6 to 8 weeks. The study is planned to enroll approximately 24 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A Hyperhidrosis Disease Severity Scale (HDSS) score of 3 or 4.
* A diagnosis of primary, axillary hyperhidrosis, defined as excessive, bilateral, axillary sweating of at least 6 months duration without apparent cause and with at least 1 of the following characteristics: subject has a positive family history of hyperhidrosis, hyperhidrosis is bilateral and relatively symmetrical, subject experienced first episode of hyperhidrosis before 25 years of age, subject experiences cessation of focal sweating during sleep.
* A baseline gravimetric assessment of at least 50 milligrams sweat produced at rest by each axilla during a period of 5 minutes (measurements can be repeated up to 2 times on two different days, screening and baseline visits, but subjects need to qualify on at least one occasion).
* Male.
* A female is eligible to enter and participate in the study if she is of:

Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, > 45 years, in the absence of hormone replacement therapy. In questionable cases for women < 60 years of age, a blood sample with simultaneous follicle stimulating hormone and estradiol falling into the central laboratory's postmenopausal reference range is confirmatory.

OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician) for the duration of the study: abstinence; oral contraceptive, either combined or progestogen alone; injectable progestogen; implants of levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device (IUD) or intrauterine system (IUS) that meets the standard operating procedure effectiveness criteria as stated in the product label; male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject; double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository

* If subjects have shaved axilla or removed hair by other means within the last 2 weeks, there should be minimal to no irritation.
* Capable of giving signed informed consent which includes compliance with the pre-specified requirements and restrictions.

Exclusion Criteria:

* Unstable or life threatening cardiac disease. In the opinion of the investigator, use should only be considered if the benefit is likely to outweigh the risk in conditions such as: myocardial infarction or unstable angina in the last 6 months, unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months, New York Heart Association (NYHA) Class IV heart failure.
* Diagnosis of narrow-angle glaucoma, urinary retention, prostatic hypertrophy or bladder neck obstruction that in the opinion of the study investigator or GlaxoSmithKline (GSK) Medical Monitor would prevent use of an anticholinergic and therefore study participation.
* Irritation or active infection of axillary area, including sweat glands.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones that the investigator deems clinically significant).
* Alanine aminotransferase (ALT) > 2 x Upper Limit of Normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) at screening.
* Corrected QT Interval (QTc) > 450 milliseconds (ms) or QTc > 480 ms in subjects with Bundle Branch Block.

The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read.

The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.

For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used.

* Prior surgical procedure for hyperhidrosis.
* Axillary treatment with radiofrequency and microwave devices.
* Treatment with axillary iontophoresis within 4 weeks prior to Baseline/Day 1.
* Menopausal women who have had symptoms of menopause such as sweating or flushing within 3 years of the study.
* Used any prohibited medication within the indicated washout period.
* Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, sympathomimetic.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen at screening.
* A positive test for Human Immunodeficiency Virus (HIV) antibody at screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time periods prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.
* Any other condition which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study (e.g., subjects with renal failure).
* Subjects with clinically significant abnormalities in laboratory values for which, according to the investigator, study participation would put the subject at undue risk.
* Abnormal findings on screening electrocardiogram (ECG) deemed clinically significant by the Investigator.
* Women who are pregnant or lactating or are planning on becoming pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (2):
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Austin, Texas
- GSK Investigational Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study conducted between 23 November 2015 to 25 February 2016. The data for population pharmacokinetic (PK) analysis was pooled from the earlier two studies including LHH117157 (NCT01934153) (6 participants from Cohort B) and AC4112008 (NCT01110018) (9 participants) with the data of the current study.
Pre-assignment Details: A total of 28 participants randomized in this study. Because of a system configuration error, randomization numbers were assigned to 5 screen failure participants. However, these participants did not enter the study and not dosed, remaining 23 participants (18- Umeclidinium; 5- Placebo) included in Full Analysis Population.
Groups:
- 202093: Umeclidinium, 2 mg/cm^2 of 1.85%, OD: Participants topically applied Umeclidinium 2 milligram per square centimeter (mg/cm^2) of the 1.85%, administered once daily (OD) to both axillae, at night before going to bed for 14 days.
- 202093: Vehicle: Participants topically applied vehicle, OD to both axillae, at night before going to bed for 14 days.
- AC4112008: GSK573719: Each participant received single dose of treatment in the following order of intravenous GSK573719 20 µg followed by oral GSK573719 1000 μg followed by intravenous GSK573719 50 µg, followed by inhaled GSK573719 1000 μg followed by intravenous GSK573719 65 µg in period 1, 2, 3, 4 and 5 respectively. The washout was of 5 days between two consecutive periods.
- LHH117157: Cohort B: A single dose of topically applied [14C] umeclidinium was administered to the occluded axilla. The dose to be administered was 165 mg of a 1.85% weight/ weight (w/w) solution umeclidinium (equivalent to a 2.2% umeclidinium bromide solution) applied to 40 centimeter squared (cm^2) surface area of occluded axilla (resulting in a calculated net amount of active umeclidinium of 3.06 mg).
Period: Overall Study
Arm/Group | 202093: Umeclidinium, 2 mg/cm^2 of 1.85%, OD | 202093: Vehicle | AC4112008: GSK573719 | LHH117157: Cohort B
Started | 18 | 5 | 10 | 6
Completed | 17 | 5 | 9 | 6
Not Completed | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 202093: Umeclidinium, 2 mg/cm^2 of 1.85%, OD: Participants topically applied Umeclidinium 2 mg/cm^2 of the 1.85% formulation, administered OD to both axillae, at night before going to bed for 14 days.
- LHH117157: Cohort B: A single dose of topically applied [14C] umeclidinium was administered to the occluded axilla. The dose to be administered was 165 mg of a 1.85% (w/w) solution umeclidinium (equivalent to a 2.2% umeclidinium bromide solution) applied to 40 (cm^2) surface area of occluded axilla (resulting in a calculated net amount of active umeclidinium of 3.06 mg).
- Total: Total of all reporting groups
Arm/Group | 202093: Umeclidinium, 2 mg/cm^2 of 1.85%, OD | 202093: Vehicle | AC4112008: GSK573719 | LHH117157: Cohort B | Total
Number analyzed (Participants) | 18 | 5 | 10 | 6 | 39
Age, Customized [Count of Participants; unit: Participants]
  19 to 64 Years | 18 | 5 | 10 | 6 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 0 | 0 | 13
  Male | 9 | 1 | 10 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 18 | 3 | 10 | 6 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Concentration After Repeat Dosing of Umeclidinium
Description: Pharmacokinetic blood sampling was done at the following time points: Day 12 (pre-dose), Day 13 (pre-dose), Day 14 (pre-dose), Day 15 (3 hours [h], 6 h, 9 h, 10 h, 12 h, 16 h, and 24 h following the Day 14 dose), Day 16 (36 h and 48 h following the Day 14 dose). Approximately 3 ml of blood was taken at each timepoint. Mean and standard deviation of the umeclidinium concentration was reported. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Day 12 to Day 16
Population: Pharmacokinetic Concentration Population defined as all participants in the Safety population for whom at least one pharmacokinetic sample was obtained and analyzed. Safety Population is defined as all participants who received at least one dose of a study drug in this study (202093)
Measure: Mean (Standard Deviation); unit: picogram per millilitre (pg/ml)
Groups:
- Umeclidinium, 2 mg/cm^2 of 1.85%, OD: Participants topically applied Umeclidinium 2 mg/cm^2 of the 1.85% formulation, administered OD to both axillae, at night before going to bed for 14 days.
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD
Number analyzed (Participants) | 18
picogram per millilitre (pg/ml)
  DAY 12, Pre-dose: number analyzed (Participants) | 12
  DAY 12, Pre-dose | 33.09 (23.206)
  DAY 13, Pre-dose: number analyzed (Participants) | 13
  DAY 13, Pre-dose | 29.86 (20.981)
  DAY 14, Pre-dose: number analyzed (Participants) | 15
  DAY 14, Pre-dose | 41.22 (42.465)
  Day 14, 3 h: number analyzed (Participants) | 16
  Day 14, 3 h | 42.72 (57.839)
  Day 14, 6 h: number analyzed (Participants) | 16
  Day 14, 6 h | 53.68 (69.157)
  Day 14, 9 h: number analyzed (Participants) | 16
  Day 14, 9 h | 57.32 (74.719)
  Day 14, 10 h: number analyzed (Participants) | 16
  Day 14, 10 h | 57.24 (77.945)
  Day 14, 12 h: number analyzed (Participants) | 15
  Day 14, 12 h | 50.72 (63.468)
  Day 14, 16 h: number analyzed (Participants) | 16
  Day 14, 16 h | 35.42 (37.727)
  Day 14, 24 h: number analyzed (Participants) | 16
  Day 14, 24 h | 31.50 (29.458)
  Day 14, 36 h: number analyzed (Participants) | 16
  Day 14, 36 h | 30.76 (46.979)
  Day 14, 48 h: number analyzed (Participants) | 16
  Day 14, 48 h | 14.28 (14.739)

2. Primary Outcome: Maximum Observed Concentration (Cmax) and Pre-dose (Trough) Concentration at the End of the Dosing Interval (Ctau) After Repeat Dosing of Umeclidinium
Description: Pharmacokinetic blood sampling was done at Day 14 (pre-dose), Day 15 (3 h, 6 h, 9 h, 10 h, 12 h, 16 h, and 24 h following the Day 14 dose), Day 16 (36 h and 48 h following the Day 14 dose). Cmax and Ctau was determined directly from the concentration-time data.
Time Frame: Day 14 (pre-dose), Day 15 (3 h, 6 h, 9 h, 10 h, 12 h, 16 h, and 24 h following the Day 14 dose), Day 16 (36 h and 48 h following the Day 14 dose)
Population: Pharmacokinetic Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD
Number analyzed (Participants) | 18
pg/mL
  Cmax, Day 14: number analyzed (Participants) | 16
  Cmax, Day 14 | 44.79 (175.27)
  Ctau, Day 12: number analyzed (Participants) | 12
  Ctau, Day 12 | 27.94 (63.30)
  Ctau, Day 13: number analyzed (Participants) | 13
  Ctau, Day 13 | 25.81 (55.40)
  Ctau, Day 14: number analyzed (Participants) | 12
  Ctau, Day 14 | 39.60 (87.68)
  Ctau, Day 15: number analyzed (Participants) | 14
  Ctau, Day 15 | 29.63 (66.76)

3. Primary Outcome: Mean Time to Reach Cmax (Tmax) of Umeclidinium After Repeat Dosing
Description: Pharmacokinetic blood sampling was done at Day 14 (pre-dose), Day 15 (3 h, 6 h, 9 h, 10 h, 12 h, 16 h, and 24 h following the Day 14 dose), Day 16 (36 h and 48 h following the Day 14 dose). Tmax was determined directly from the concentration-time data.
Time Frame: Day 14 to Day 16
Population: Pharmacokinetic Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD
Number analyzed (Participants) | 14
h | 10.25 (7.985)

4. Primary Outcome: Mean Terminal Plasma Elimination Rate Constant (Lambda Z) of Umeclidinium After Repeat Dosing
Description: Pharmacokinetic blood sampling was done at Day 14 (pre-dose), Day 15 (3 h, 6 h, 9 h, 10 h, 12 h, 16 h, and 24 h following the Day 14 dose), Day 16 (36 h and 48 h following the Day 14 dose). Derivation of lambda-Z was planned. However, the parameter could not be derived for any of the participant included in the study because of insufficient data in the elimination phase (< 3 data points, coefficient of determination (R^2) was not adequate).
Time Frame: Day 14 to Day 16
Population: Pharmacokinetic Concentration Population
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD
Number analyzed (Participants) | 0

5. Primary Outcome: Terminal Phase Half-life (t1/2) of Umeclidinium After Repeat Dosing
Description: Pharmacokinetic blood sampling was done at Day 14 (pre-dose), Day 15 (3 h, 6 h, 9 h, 10 h, 12 h, 16 h, and 24 h following the Day 14 dose), Day 16 (36 h and 48 h following the Day 14 dose). Derivation of t1/2 was planned. However, the parameter could not be derived for any of the participant included in the study because of insufficient data in the elimination phase (< 3 data points, coefficient of determination (R^2) was not adequate).
Time Frame: Day 14 to Day 16
Population: Pharmacokinetic Concentration Population
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD
Number analyzed (Participants) | 0

6. Primary Outcome: Mean Area Under the Concentration-time Curve (AUC) From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Across All Treatments (0-t) and AUC Over the Dosing Interval (0-tau) of Umeclidinium After Repeat Dosing
Description: Pharmacokinetic blood sampling was done at Day 14 (pre-dose), Day 15 (3 h, 6 h, 9 h, 10 h, 12 h, 16 h, and 24 h following the Day 14 dose), Day 16 (36 h and 48 h following the Day 14 dose). Calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. Geometric mean of log-transformed values of AUC were reported.
Time Frame: Day 14 to Day 16
Population: Pharmacokinetic Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD
Number analyzed (Participants) | 16
h*pg/mL
  AUC(0-t) | 1036.90 (142.63)
  AUC(0-tau) | 703.67 (108.61)

7. Primary Outcome: Composite Population Pharmacokinetics Parameter: Volume of Distribution in Central Compartment (V1) and Volume of Distribution in Peripheral Compartment (V2)
Description: Pharmacokinetic blood sampling was done at Pre-dose, 3h, 6h, 9h, 10h, 12h, 16h, 24h, 36h, 48h of current study (202093), pre-dose, 10, 20, 30, 32, 35, 45 minute, 1h, 2h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h for study AC4112008, and Pre-dose, 2h, 4h, 5h, 6h, 8h, 8.5h, 9h, 9.5h, 10h, 11h, 12h, 13h, 14h, 16h, 24h, 30h, 36h, 48h, 72h for study number LHH117157. Plasma umeclidinium concentration time data following administration to axilae of hyperhidrosis participants from the current study (202093) were pooled with data from the occluded axilla cohort from study LHH117157 and the IV infusion data from study AC4112008 in order modify the existing population PK model for dermal umeclidinium. Plasma concentration-time data was subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK model. The data for V1 and V2 was reported as mean (estimate) with relative standard error (RSE). RSE= (Standard error of the estimate/ Final parameter estimate) X 100.
Time Frame: Day 12 to Day 16
Population: Pharmacokinetic Concentration Populations from studies 202093 (16 participants), AC4112008 (9 participants) and LHH117157 (6 participants) were pooled to population Pk parameter analysis.
Measure: Mean (Standard Error); unit: Litre (L)
Groups:
- Pooled Umeclidinium Population PK Arm: This arm is consisted of pooled PK populations from study 202093, AC4112008 and LHH117157. In the study 202093 participants topically applied Umeclidinium 2 mg/cm^2 of 1.85%, administered OD to both axillae, at night before going to bed for 14 days. In the study AC411200 each participant received single dose of treatment in the following of order intravenous GSK573719 20 µg followed by oral GSK573719 1000 μg followed by intravenous GSK573719 50 µg, followed by inhaled GSK573719 1000 μg followed by intravenous GSK573719 65 µg in period 1, 2, 3, 4 and 5 respectively. Washout was of 5 days between two consecutive periods. In the study LHH117157 a single dose of topically applied [14C] umeclidinium was administered to the occluded axilla. The dose to be administered was 165 mg of a 1.85% w/w solution umeclidinium (equivalent to a 2.2% umeclidinium bromide solution) applied to 40 cm^2 surface area of occluded axilla (resulting in a calculated net amount of active umeclidinium of 3.06 mg)
Arm/Group | Pooled Umeclidinium Population PK Arm
Number analyzed (Participants) | 31
Litre (L)
  V1 | 7.44 (9.65)
  V2 | 333 (22.6)

8. Primary Outcome: Composite Population Pharmacokinetics Parameter: Elimination Clearance (CL) and Inter-compartmental Clearance (Q)
Description: Pharmacokinetic blood sampling was done at Pre-dose, 3h, 6h, 9h, 10h, 12h, 16h, 24h, 36h, 48h of current study (202093), pre-dose, 10, 20, 30, 32, 35, 45 minute, 1h, 2h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h for study AC4112008, and Pre-dose, 2h, 4h, 5h, 6h, 8h, 8.5h, 9h, 9.5h, 10h, 11h, 12h, 13h, 14h, 16h, 24h, 30h, 36h, 48h, 72h for study number LHH117157. Plasma umeclidinium concentration time data following administration to axilae of hyperhidrosis participants from the current study (202093) were pooled with data from the occluded axilla cohort from study LHH117157 and the IV infusion data from study AC4112008 in order modify the existing population PK model for dermal umeclidinium. Plasma concentration-time data was subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK model. The data for CL and Q was reported as mean (estimate) with RSE. RSE= (Standard error of the estimate/ Final parameter estimate) X 100.
Time Frame: Day 12 to Day 16
Population: as for outcome 7
Measure: Mean (Standard Error); unit: L/h
Arm/Group | Pooled Umeclidinium Population PK Arm
Number analyzed (Participants) | 31
L/h
  CL | 53.2 (11.1)
  Q | 43.1 (24.6)

9. Primary Outcome: Composite Population Pharmacokinetics Parameter: Absorption Rate Constant (Ka)
Description: Pharmacokinetic blood sampling was done at Pre-dose, 3h, 6h, 9h, 10h, 12h, 16h, 24h, 36h, 48h of current study (202093), pre-dose, 10, 20, 30, 32, 35, 45 minute, 1h, 2h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h for study AC4112008, and Pre-dose, 2h, 4h, 5h, 6h, 8h, 8.5h, 9h, 9.5h, 10h, 11h, 12h, 13h, 14h, 16h, 24h, 30h, 36h, 48h, 72h for study number LHH117157. Plasma umeclidinium concentration time data following administration to axilae of hyperhidrosis participants from the current study (202093) were pooled with data from the occluded axilla cohort from study LHH117157 and the IV infusion data from study AC4112008 in order modify the existing population PK model for dermal umeclidinium. Plasma concentration-time data was subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK model. The data for Ka was reported as mean (estimate) with RSE. RSE= (Standard error of the estimate/ Final parameter estimate) X 100.
Time Frame: Day 12 to Day 16
Population: as for outcome 7
Measure: Mean (Standard Error); unit: 1/h
Arm/Group | Pooled Umeclidinium Population PK Arm
Number analyzed (Participants) | 31
1/h | 0.012 (48.6)

10. Primary Outcome: Composite Population Pharmacokinetics Parameter: Absolute Plasma Bioavailability Following Administration to Axilae (FA) Fraction of the Bioavailable Drug Absorbed Through a Zero Order Process (F2 [FIXED])
Description: Pharmacokinetic blood sampling was done at Pre-dose, 3h, 6h, 9h, 10h, 12h, 16h, 24h, 36h, 48h of current study (202093), pre-dose, 10, 20, 30, 32, 35, 45 minute, 1h, 2h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h for study AC4112008, and Pre-dose, 2h, 4h, 5h, 6h, 8h, 8.5h, 9h, 9.5h, 10h, 11h, 12h, 13h, 14h, 16h, 24h, 30h, 36h, 48h, 72h for study number LHH117157. Plasma umeclidinium concentration time data following administration to axilae of hyperhidrosis participants from the current study (202093) were pooled with data from the occluded axilla cohort from study LHH117157 and the IV infusion data from study AC4112008 in order modify the existing population PK model for dermal umeclidinium. Plasma concentration-time data was subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK model. The data for FA and F2 (FIXED) was reported as mean (estimate) with RSE. RSE= (Standard error of the estimate/ Final parameter estimate) x 100.
Time Frame: Day 12 to Day 16
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Pooled Umeclidinium Population PK Arm
Number analyzed (Participants) | 31
Ratio
  FA | -5.05 (3.15)
  F2 | -2 (0)

11. Primary Outcome: Composite Population Pharmacokinetics Parameter: Duration of the Zero Order Process and Lag Time for the First Order Absorption Process (ALAG1)
Description: Pharmacokinetic blood sampling was done at Pre-dose, 3h, 6h, 9h, 10h, 12h, 16h, 24h, 36h, 48h of current study (202093), pre-dose, 10, 20, 30, 32, 35, 45 minute, 1h, 2h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h for study AC4112008, and Pre-dose, 2h, 4h, 5h, 6h, 8h, 8.5h, 9h, 9.5h, 10h, 11h, 12h, 13h, 14h, 16h, 24h, 30h, 36h, 48h, 72h for study number LHH117157. Plasma umeclidinium concentration time data following administration to axilae of hyperhidrosis participants from the current study (202093) were pooled with data from the occluded axilla cohort from study LHH117157 and the IV infusion data from study AC4112008 in order modify the existing population PK model for dermal umeclidinium. Plasma concentration-time data was subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK model. The data for ALAG1 was reported as mean (estimate) with RSE. RSE= (Standard error of the estimate/ Final parameter estimate) x 100.
Time Frame: Day 12 to Day 16
Population: as for outcome 7
Measure: Mean (Standard Error); unit: h
Arm/Group | Pooled Umeclidinium Population PK Arm
Number analyzed (Participants) | 31
h | 2.56 (26.5)

12. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Event (SAE)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Over a period of 28 days
Population: Safety population of study number 202093, LHH117157 (Cohort B) and AC4112008 were used to report AEs.
Measure: Count of Participants; unit: Participants
Groups:
- Vehicle: Participants topically applied vehicle, OD to both axillae, at night before going to bed for 14 days.
- AC4112008: GSK573719: Each participants received single dose of treatment in the following order intravenous GSK573719 20 µg followed by oral GSK573719 1000 μg followed by intravenous GSK573719 50 µg, followed by inhaled GSK573719 1000 μg followed by intravenous GSK573719 65 µg in period 1, 2, 3, 4 and 5 respectively. The washout was of 5 days between two consecutive periods.
- LHH117157: Cohort B: A single dose of topically applied [14C] umeclidinium administered to the occluded axilla. The dose to be administered was 165 mg of a 1.85% (w/w) solution Umeclidinium (equivalent to a 2.2% Umeclidinium bromide solution) applied to 40 (cm^2) surface area of occluded axilla (resulting in a calculated net amount of active Umeclidinium of 3.06 mg).
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle | AC4112008: GSK573719 | LHH117157: Cohort B
Number analyzed (Participants) | 18 | 5 | 10 | 6
Participants
  Any AE | 9 | 2 | 6 | 2
  Any SAE | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Abnormal Values of Potential Clinical for Electrocardiogram (ECG)
Description: Single 12-lead ECGs was obtained at Day 1, Day 14 and Day 28 during the study. The standard ECG criteria of potential clinical importance were 1) absolute QTc Interval, > 450 milliseconds (msec), 2) absolute PR Interval, <110 msec, 3) absolute QRS Interval, < 75 msec and 4) increase from baseline in QTc > 60 msec. The number of participants with potentially clinically significant ECG findings at any visit were reported.
Time Frame: Up to Day 28
Population: Safety Population is defined as all participants who received at least one dose of a study drug in this study (202093).
Measure: Count of Participants; unit: Participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 18 | 5
Participants
  Low QRS | 3 | 0
  High QRS | 2 | 0
  High QTcB | 1 | 1
  Low PR interval | 0 | 1

14. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance at Any Time on Treatment
Description: The clinical chemistry parameters analyzed were albumin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, bicarbonate, blood urea nitrogen, calcium, chloride, creatinine, gamma glutamyl transferase, glucose, potassium, sodium, total and direct bilirubin, total protein, uric acid. Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important clinical chemistry findings at any visit were reported.
Time Frame: Up to day 28
Population: Safety Population is defined as all participants who received at least one dose of a study drug in this study (202093).
Measure: Count of Participants; unit: Participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 18 | 5
Participants
  High, alanine aminotransferase | 1 | 1
  High, aspartate aminotransferase | 1 | 1
  High, glucose | 1 | 1

15. Primary Outcome: Number of Participants With Clinical Hematology Abnormalities of Potential Clinical Importance at Any Time on Treatment.
Description: The hematology parameters analyzed were basophils, eosinophils, erythrocyte mean corpuscular hemoglobin concentration, erythrocyte mean corpuscular hemoglobin, erythrocyte mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, monocytes, neutrophils, platelets, and reticulocytes. Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important hematology findings at any visit were reported.
Time Frame: Up to Day 28
Population: Safety Population is defined as all participants who received at least one dose of a study drug in this study (202093).
Measure: Count of Participants; unit: Participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 18 | 5
Participants
  Low, Neutrophils | 1 | 0
  High, Hematocrit | 1 | 0

16. Primary Outcome: Number of Participants With Urinalysis Abnormalities of Potential Clinical Importance at Any Time on Treatment
Description: The urinalysis parameters analyzed were specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination. Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important urinalysis findings at any visit were reported.
Time Frame: Up to Day 28
Population: Safety Population is defined as all participants who received at least one dose of a study drug in this study (202093).
Measure: Count of Participants; unit: Participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 18 | 5
Participants | 1 | 0

17. Primary Outcome: Number of Participants With Abnormal Values of Potential Clinical for Vital Signs
Description: The potential clinical importance ranges (low and high) of the vital sign parameters were for systolic blood pressure (<85 and >160 millimeter of mercury [mmHg]), diastolic blood pressure (<45 and >100 mmHg) and heart rate (<40 and >110 beats per minute). Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important vital parameter findings at any visit were reported.
Time Frame: Up to 28 days
Population: Safety Population is defined as all participants who received at least one dose of a study drug in this study (202093).
Measure: Count of Participants; unit: Participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 18 | 5
Participants | 1 | 0

18. Primary Outcome: Number of Participants With Local Tolerability Assessment Score Over 28 Days
Description: The investigator or designated evaluator assessed skin tolerability at each visit using the 5-point tolerability scale. Tolerability of the topical application was assessed and scored as, 0- none (no evidence of local intolerance), 1-mild (minimal erythema and/or edema, slight glazed appearance), 2-moderate (definite erythema and/or edema with peeling and/or cracking but needs no adaptation of posology), 3-severe (erythema, edema glazing with fissures, few vesicles or papules), 4- very severe (strong reaction spreading beyond the treated area, bullous reaction, erosions).
Time Frame: Days 1, 2, 4, 5, 6, 7, 8, 9, 10, 13, 14, 15, 16, and 23
Population: Safety Population is defined as all participants who received at least one dose of a study drug in this study (202093).
Measure: Count of Participants; unit: Participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 18 | 5
Participants
  Day 1, Mild, n= 18, 5 | 2 | 0
  Day 2, Mild, n= 18, 5 | 2 | 2
  Day 4, Moderate, n= 18, 5 | 1 | 0
  Day 5, Mild, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 5, Mild, n= 17, 5 | 2 | 0
  Day 6, Mild, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 6, Mild, n= 17, 5 | 2 | 1
  Day 7, Mild, n= 18, 5 | 2 | 0
  Day 8, Mild, n= 15, 5: number analyzed (Participants) | 15 | 5
  Day 8, Mild, n= 15, 5 | 3 | 0
  Day 9, Mild, n= 16, 5: number analyzed (Participants) | 16 | 5
  Day 9, Mild, n= 16, 5 | 1 | 0
  Day 10, Mild, n= 16, 5: number analyzed (Participants) | 16 | 5
  Day 10, Mild, n= 16, 5 | 0 | 1
  Day 13, Mild, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 13, Mild, n= 17, 5 | 2 | 1
  Day 13, Moderate, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 13, Moderate, n= 17, 5 | 1 | 0
  Day 14, Mild, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 14, Mild, n= 17, 5 | 2 | 0
  Day 15, Mild, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 15, Mild, n= 17, 5 | 1 | 0
  Day 16, Mild, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 16, Mild, n= 17, 5 | 1 | 1
  Day 23, Mild, n= 17, 5: number analyzed (Participants) | 17 | 5
  Day 23, Mild, n= 17, 5 | 2 | 0

19. Secondary Outcome: Change From Baseline in Amount of Sweat Produced at Day 15
Description: Amount of sweat produced was determined by gravimetry analysis for axilla. Filter paper in a sealed container was weighed. After drying the axillary surface, the filter paper was removed from the container and applied to the axilla. The paper was covered with plastic wrap and tape around the edges with paper tape. The filter paper was left in contact with the axilla for a period of 5 minutes as measured by a stopwatch. The filter paper was then replaced in the sealed container and re-weighed. Rate of sweat production was calculated in milligrams/minute (mg/min). Participants remained at rest for 20-30 minute before the measurements in order to reduce external interference. Measurements were carried out in a climate-controlled environment (21-24°C). Assessments conducted at Day 1, Pre-dose time point (average pre-dose measurements for both left and right measurements) were considered as Baseline values. Change from baseline was calculated as Day 15 value minus Baseline value.
Time Frame: Baseline (Pre-dose, Day 1) and Day 15
Population: Full Analysis population comprised of participants receiving study medication and having at least 1 post baseline visit. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/ min
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 17 | 5
mg/ min | -0.0571 (0.09402) | -0.0164 (0.01735)

20. Secondary Outcome: Percentage of Participants With Cut-points for Percent Change From Baseline in Sweat Production at Day 15
Description: Amount of sweat produced was determined by gravimetry analysis for axilla. Filter paper in a sealed container was weighed. After drying the axillary surface, the filter paper was removed from the container and applied to the axilla. The paper was covered with plastic wrap and tape around the edges with paper tape. The filter paper was left in contact with the axilla for a period of 5 minutes as measured by a stopwatch. The filter paper was then replaced in the sealed container and re-weighed. Rate of sweat production was calculated in milligrams/minute. Assessments conducted at Day 1, Pre-dose time point (average pre-dose measurements for both left and right measurements) were considered as Baseline values. Percent change from Baseline= 100 x ( Day 15 value - Baseline value) / Baseline value. The percentage of participants with cutpoints (-30%, -50, -75%) for percent change from Baseline in sweat production were presented.
Time Frame: Baseline (Pre-dose, Day 1) and Day 15
Population: Full Analysis population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 18 | 5
Percentage of participants
  <=-30% | 59 | 60
  <=-50% | 41 | 40
  <=-75% | 29 | 20
Statistical Analysis 1: Comparison: Umeclidinium, 2 mg/cm^2 of 1.85%, OD vs Vehicle; Umeclidinium, 2 mg/cm^2 of 1.85%, OD Vs Vehicle: <=-30%; Test type: Superiority or Other; Percent difference in treatment = -1, 95% CI 2-sided [-42.2 to 39.9]
Statistical Analysis 2: Comparison: Umeclidinium, 2 mg/cm^2 of 1.85%, OD vs Vehicle; Umeclidinium, 2 mg/cm^2 of 1.85%, OD vs Vehicle: <=-50%; Test type: Superiority or Other; Percent difference in treatment = 1, 95% CI 2-sided [-39.9 to 42.2]
Statistical Analysis 3: Comparison: Umeclidinium, 2 mg/cm^2 of 1.85%, OD vs Vehicle; Umeclidinium, 2 mg/cm^2 of 1.85%, OD Vs Vehicle: <=-70%; Test type: Superiority or Other; Percent difference in treatment = 9, 95% CI 2-sided [-25.2 to 44.0]

21. Secondary Outcome: Change in Hyperhidrosis Disease Severity Scale (HDSS) at Day 15
Description: The HDSS is a 4-point scale which used to assess the impact of disease. The scores were define as, 1- My (underarm) sweating is never noticeable and never interferes with my daily Activities; 2- My (underarm) sweating is tolerable but sometimes interferes with my daily activities; 3- My (underarm) sweating is barely tolerable and frequently interferes with my daily activities; 4- My (underarm) sweating is intolerable and always interferes with my daily activities. Average score of both left and right underarms were used for analysis. The possible average score range from 1 (minimum) to 4 (maximum). The reduction in score on the scale presents betterment and increase in the score represents worsening. Assessments conducted at Day 1, pre-dose time point (average pre-dose measurements for both left and right underarm measurements) were considered as Baseline values. Change from baseline was calculated as Day 15 Visit Value minus Baseline values.
Time Frame: Baseline (Pre-dose, Day 1) and Day 15
Population: Full Analysis population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Error); unit: Score on Scale
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 17 | 5
Score on Scale | -1.4 (1.00) | -0.6 (0.89)

22. Secondary Outcome: Percentage of Participants With 2-point Decrease From Baseline to Day 15 in HDSS Score
Description: HDSS is a 4-point scale which used to assess the impact of disease. The scores are define as, 1- My (underarm) sweating is never noticeable and never interferes with my daily Activities; 2- My (underarm) sweating is tolerable but sometimes interferes with my daily activities; 3- My (underarm) sweating is barely tolerable and frequently interferes with my daily activities; 4- My (underarm) sweating is intolerable and always interferes with my daily activities. Average score of both left and right underarms were used for analysis. The possible average score range from 1 (minimum) to 4 (maximum). Increase in score on scale represents worsening. Assessments conducted at Day 1, pre-dose time point (average pre-dose measurements for both left and right underarm measurements) were considered as Baseline values. Change from baseline was calculated as Day 15 Visit Value minus Baseline values. Percentage of participants with 2-point decrease from Baseline to Day 15 in HDSS score were reported.
Time Frame: Baseline (Pre-dose, Day 1) and Day 15
Population: Full Analysis population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Umeclidinium, 2 mg/cm^2 of 1.85%, OD | Vehicle
Number analyzed (Participants) | 17 | 5
Percentage of participants | 47 | 20
Statistical Analysis 1: Comparison: Umeclidinium, 2 mg/cm^2 of 1.85%, OD vs Vehicle; Test type: Superiority or Other; Percent difference in treatment = 27, 95% CI 2-sided [-8.5 to 62.6]

ADVERSE EVENTS:
Time Frame: AEs were collected up to end of the follow-up. The end of the follow-up duration for the study 202093 was Day 28, for the study AC4112008 was Day 50 and for the study LHH117157 Day 18.
Description: Safety population of study number 202093, LHH117157 (Cohort B) and AC4112008 were used to report SAEs and nSAEs.
Groups:
- 202093:Umeclidinium: Participants topically applied Umeclidinium 2 mg/cm^2 of the 1.85% formulation, administered OD to both axillae, at night before going to bed for 14 days.
- 202093:Vehicle: Participants topically applied vehicle, OD to both axillae, at night before going to bed for 14 days.
Arm/Group | 202093:Umeclidinium | 202093:Vehicle | AC4112008: GSK573719 | LHH117157: Cohort B
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/5 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/5 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 9/18 | 2/5 | 6/10 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 202093:Umeclidinium (N=18) | 202093:Vehicle (N=5) | AC4112008: GSK573719 (N=10) | LHH117157: Cohort B (N=6)
Application site pain (General disorders) | 3 | 0 | 0 | 0 — General disorders and administration site conditions
Application site pruritus (General disorders) | 2 | 0 | 0 | 0 — General disorders and administration site conditions
Application site erythema (General disorders) | 1 | 0 | 0 | 0 — General disorders and administration site conditions
Application site exfoliation (General disorders) | 1 | 0 | 0 | 0 — General disorders and administration site conditions
Application site paraesthesia (General disorders) | 0 | 1 | 0 | 0 — General disorders and administration site conditions
Chest pain (General disorders) | 1 | 0 | 0 | 0 — General disorders and administration site conditions
Headache (Nervous system disorders) | 4 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 (0) | 0 | 2 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Application site iiritation (General disorders) | 0 | 0 | 0 | 1
Application site dryness (General disorders) | 0 | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pain in extrmity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.